CLINICAL TRIAL: NCT03187340
Title: Monitored Breathing Awareness Therapy for Insomnia Disorder in Older Adults: Randomized Study
Brief Title: Monitored Breathing Awareness Therapy for Insomnia Disorder in Older Adults-2
Acronym: MBAT-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nalaka Gooneratne (Other)
Collaborators: Advanced Medical Electronics (Other)
Responsible Party: Sponsor-Investigator, Nalaka Gooneratne, Associate Professor, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10053582
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep education and relaxation 1 (Active Comparator): Behavioral education intervention about sleep and relaxation
  Interventions: Behavioral: Sleep education and relaxation 1
- Sleep education and relaxation 2 (Experimental): Behavioral education intervention about sleep and relaxation
  Interventions: Behavioral: Sleep education and relaxation 2

INTERVENTIONS:
Behavioral: Sleep education and relaxation 1 — Sleep hygiene and relaxation training; Sleep education and relaxation 1
  Arms: Sleep education and relaxation 1
Behavioral: Sleep education and relaxation 2 — Modified sleep hygiene and relaxation training; Sleep education and relaxation 2
  Arms: Sleep education and relaxation 2

SUMMARY:
Insomnia can be a chronic problem that leads to significant daytime fatigue, stress and numerous negative health consequences including depression. Advanced Medical Electronics, in partnership with researchers are the University of Pennsylvania, propose developing an innovative, non-drug, low-risk, intervention that can be implemented on mobile devices for the treatment of insomnia

ELIGIBILITY:
Inclusion Criteria: 1) Sleep onset latency > 30 min for at least 3 nights per week

Exclusion Criteria: 1) Unable to perform tests due to inability to communicate verbally/blindness, inability to write and read in English (the study questionnaires are in English and do not exist in validated form for other languages). 2) Cognitive impairment; cognitively impaired patients may not be able to comply with the protocol). 3) History of a diagnosed non-insomnia sleep disorder, such as sleep apnea or circadian rhythm disorder 4) Upper extremity motor impairment that would preclude MBAT therapy (e.g., quadriplegia).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep onset latency | four weeks
  time to fall asleep

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
At conclusion of study as per NIH guidelines